CLINICAL TRIAL: NCT06714474
Title: Effectiveness of Virtual Simulation Game in Teaching Venous Blood Sampling Skills to Nursing Students: a Randomized Controlled Trial
Brief Title: Effectiveness of Virtual Simulation Game in Teaching Venous Blood Sampling Skills to Nursing Students
Acronym: VSG-Venous
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinop University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); Ege University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SINOPU-HEM-RK-01
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Nursing Skill; Game-Based Learning; Students, Nursing; Gamification; Blood Sampling Procedure
Keywords: Nursing Education; Virtual Simulation Game; Nursing Students; Venous Blood Sampling

STUDY DESIGN:
Intervention Model Description: Model Description
  In this randomized controlled trial, participants are assigned to one of two parallel groups:
  Experimental Group: Participants receive training using a Virtual Simulation Game (VSG) for venous blood sampling (VBS) skills.
  Control Group: Participants receive traditional training methods for VBS skills.
  The interventions are applied concurrently, and the outcomes (knowledge, skill performance, satisfaction, confidence, and comfort) are compared between the two groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking Description In this study, outcomes assessors are blinded to the group assignments to reduce bias in evaluating participants' performance, satisfaction, confidence, and comfort levels. Participants and care providers are not blinded due to the nature of the interventions, as the experimental group engages with a Virtual Simulation Game (VSG) platform that is distinguishable from the standard teaching method used in the control group.
  No other parties are masked in this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Simulation Game Group (Experimental): Participants in this arm will receive traditional training on venous blood sampling (VBS), including theoretical instruction and hands-on practice in a laboratory setting. Additionally, they will use a Virtual Simulation Game (VSG) platform (http://www.hemsirelab.com) to enhance their learning through interactive, scenario-based training. After logging into the VSG platform with unique credentials, participants will complete the training scenarios to refine their skills before performing the procedure on peers under supervision.
  Interventions: Other: Virtual Simulation Game; Other: Traditional Training
- Traditional Education Group (Active Comparator): Participants in this arm will receive traditional training on venous blood sampling (VBS) in a laboratory setting. They will observe demonstrations and practice the procedure on peers without the use of virtual simulation
  Interventions: Other: Traditional Training

INTERVENTIONS:
Other: Virtual Simulation Game — The Virtual Simulation Game (VSG) is an interactive, scenario-based digital training tool designed to enhance venous blood sampling (VBS) skills. Participants engage with the VSG platform to complete modules that simulate real-life clinical scenarios, allowing them to refine decision-making and procedural skills in a safe, controlled environment. This intervention is used in addition to traditional training to reinforce learning through repetition and feedback.
  Arms: Virtual Simulation Game Group
Other: Traditional Training — Traditional training consists of theoretical instruction and hands-on practice sessions conducted in a laboratory setting. Participants observe VBS demonstrations, followed by supervised practice on peers to develop their procedural skills. This intervention represents the standard educational approach for VBS and serves as the comparator in this study.

SUMMARY:
The goal of this randomized controlled trial is to evaluate the effectiveness of the Virtual Simulation Game (VSG) method in teaching venous blood sampling (VBS) skills to second-year nursing students. The study aims to provide a safe, engaging, and innovative learning environment for nursing students, enabling them to improve their skills without compromising patient safety.

The main questions the study seeks to answer are:

Does VSG training improve nursing students' knowledge levels in VBS education? Does VSG training enhance nursing students' practical performance in VBS procedures? Does VSG training increase nursing students' satisfaction with VBS education? Does VSG training boost nursing students' confidence in performing VBS? Does VSG training enhance nursing students' comfort during VBS practice? Researchers will compare the Virtual Simulation Game (VSG) method to the standard technique. In the VSG group, students will engage with an interactive simulation game to practice VBS skills virtually before applying them in a clinical setting. In the control group, students will practice VBS skills using traditional methods in a laboratory environment.

Participants' Tasks:

Students in the VSG group will:

Log in to the simulation platform with their credentials. Complete interactive training scenarios that mimic real-life challenges in venous blood sampling.

Practice the procedure on their peers under supervision.

Students in the control group will:

Practice VBS directly on their peers under supervision without using simulation.

After practicing, all students will be observed for 15 minutes by expert nurses for potential complications or discomfort. If needed, participants will receive medical care.

This study adheres to the CONSORT guidelines for randomized controlled trials and incorporates validated instruments to measure knowledge, skill performance, satisfaction, confidence, and comfort levels among participants. The findings aim to bridge the gap in nursing education by introducing an innovative, technology-driven approach to skill training.

DETAILED DESCRIPTION:
Simulation-based learning is essential in nursing education, especially for improving clinical decision-making and procedural skills in a risk-free environment. Virtual Simulation Games (VSGs), a form of digital learning environment, provide students with an opportunity to practice clinical scenarios in a professional role using a game-like structure. VSGs enable students to repeatedly attempt tasks, receive immediate feedback, and experience the consequences of their actions without compromising patient safety (Luctkar-Flude et al., 2021). Despite the widespread use of simulation-based training, there is a significant gap in the literature regarding the application of VSGs for fundamental nursing skills, such as venous blood sampling. Most previous studies have focused on simulations involving mannequins, and experimental designs evaluating human-based outcomes are scarce (Verkuyl et al., 2022; Keys et al., 2020).

The use of venous blood sampling procedures is a core part of healthcare services, yet errors in the process remain a significant issue. Preanalytical errors, which include hemolyzed samples, insufficient blood volume, and mislabeled samples, account for the majority (46-68%) of laboratory errors (Hammerling, 2012). These errors are preventable and often result from improper training or lack of adherence to standard protocols (Plebani, 2010). Preanalytical errors have a direct impact on patient safety, diagnostic delays, increased costs, and excessive resource use (Alcantara et al., 2022). For instance, studies have shown the average cost of a preanalytical error is $337.05 in outpatient care in the United States, while in Europe, it averages €107.62 (Green, 2013).

The training offered by this study aims to equip nursing students with practical skills to minimize such errors, emphasizing adherence to standard procedures and effective patient care practices. By combining traditional training with a VSG, this study offers a novel approach to improving education outcomes while addressing a critical need in healthcare education.

This study is a randomized controlled trial designed to assess the effectiveness of the Virtual Simulation Game (VSG) method in teaching venous blood sampling (VBS) skills to second-year nursing students. The trial uses a structured methodology to evaluate the impact of this innovative teaching tool on students' knowledge, practical skills, satisfaction, confidence, and comfort levels compared to the traditional teaching method.

Background and Rationale

Venous blood sampling is a routine yet critical procedure in healthcare, often prone to preanalytical errors that can impact patient safety and increase healthcare costs. Traditional methods of teaching VBS in nursing education focus on hands-on practice in laboratory settings, which may not adequately address the complexity of real-world challenges. The integration of virtual simulation games offers an innovative solution by providing an immersive, interactive, and repeatable environment for skill acquisition without compromising patient safety.

The Virtual Simulation Game (VSG) aligns with experiential learning theories, such as David Kolb's model, to provide nursing students with an engaging educational experience. By simulating real-life clinical scenarios, the VSG allows students to practice decision-making, receive instant feedback, and refine their skills in a low-risk environment.

Study Design

Type of Study: Randomized Controlled Trial Blinding: Single-blind (participants are aware of their assigned intervention; evaluators are blinded) Population: Second-year nursing students enrolled in the "Fundamentals of Nursing" course, who meet the inclusion criteria.

Sample Size: A total of 220 participants, with 110 students randomized to the experimental group (VSG) and 110 to the control group (traditional teaching).

Interventions

Experimental Group (VSG):

Students access the VSG platform using unique credentials. The platform includes interactive scenarios designed to mimic real-life challenges in venous blood sampling.

Students perform VBS procedures on peers after completing the virtual simulation training.

Control Group (Traditional Method):

Students receive standard instruction and practice VBS on peers in a laboratory setting.

The procedure follows conventional teaching methods without the use of virtual simulation.

Objectives

To evaluate the impact of the VSG method on nursing students' cognitive and psychomotor skills in VBS.

To assess the influence of VSG on student satisfaction, confidence, and comfort levels during VBS education.

To compare the effectiveness of VSG with the standard teaching method in reducing preanalytical errors during VBS procedures.

Hypotheses

VSG training will improve students' knowledge levels in VBS compared to traditional teaching.

VSG training will enhance students' practical performance in VBS procedures. VSG training will increase students' satisfaction with their educational experience.

VSG training will boost students' confidence in performing VBS. VSG training will improve students' comfort levels during VBS practice. Outcome Measures

Primary and secondary outcome measures include:

Primary Outcomes:

Knowledge improvement assessed using a validated questionnaire. Skill performance evaluated through a structured checklist.

Secondary Outcomes:

Student satisfaction measured using the Student Satisfaction and Self-Confidence in Learning Scale.

Confidence and comfort levels assessed via visual analog scales. Procedures

Randomization: Students will be randomized into experimental or control groups using a computer-generated sequence.

Training:

Both groups will receive a 45-minute theoretical lecture on VBS principles. The experimental group will complete VSG training before practicing on peers. The control group will directly practice on peers after the lecture.

Assessment:

Pre- and post-intervention evaluations will be conducted to measure knowledge, skill performance, satisfaction, confidence, and comfort.

Observations will be made for complications or adverse events during the practice.

Data Collection and Analysis

Data will be collected using structured forms, checklists, and validated scales. Statistical analyses will be performed using IBM SPSS Statistics, with tests including ANOVA, Kruskal-Wallis, and correlation analyses to evaluate differences and relationships between outcomes across groups.

Ethical Considerations

The study protocol has been approved by the ethics committee of Ege University Nursing Faculty.

Informed consent will be obtained from all participants. The study adheres to the Declaration of Helsinki and relevant guidelines for ethical research involving human subjects.

Significance and Innovation

The results of this study are expected to provide evidence supporting the integration of virtual simulation games into nursing curricula. This method offers a scalable and sustainable approach to enhancing nursing education, with potential benefits for improving patient safety and reducing healthcare costs through better-prepared healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

Enrolled in the "Principles and Applications in Nursing" course, specifically the "Fundamentals of Nursing Care" module, for the first time.

No prior clinical experience. No prior experience with venous blood sampling. No prior education in health sciences (e.g., not a graduate of a vocational health school or a health-related associate degree program).

Willing to voluntarily participate in the study.

Exclusion Criteria:

Diagnosed with a chronic illness, bleeding disorder, or psychiatric condition. Pregnant students. Students who have not received Hepatitis A or Hepatitis B vaccines. Students who fail to complete the study data collection forms. Students who withdraw their consent to participate during the study. Students who are absent at any stage of the study process. Students who do not complete the simulation training sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Venous Blood Sampling Knowledge Form | Pre-intervention (baseline) and post-intervention (immediately after training).
  Change in participants' knowledge of venous blood sampling procedures, assessed via a validated questionnaire.
Venous Blood Sampling Application Checklist | Pre-intervention (baseline) and post-intervention (immediately after training).
  Evaluation of participants' practical skills in venous blood sampling using a structured observational checklist.

SECONDARY OUTCOMES:
Student Satisfaction and Self-Confidence in Learning Scale | Pre-intervention (baseline) and post-intervention (immediately after training).
  Participant satisfaction with the educational experience, measured using the "Student Satisfaction and Self-Confidence in Learning Scale."
Visual Comparison (Comfort) Scale | Pre-intervention (baseline) and post-intervention (immediately after training).
  Measurement of comfort levels during venous blood sampling training using the "Visual Comparison Scale."

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Nursing Simulation Laboratory, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 01.01.2025 - 01.02.2025
Access Criteria: A signed data sharing agreement ensuring data confidentiality and adherence to ethical standards.

REFERENCES:
- [Background] Plebani M. Errors in clinical laboratories or errors in laboratory medicine? Clin Chem Lab Med. 2006;44(6):750-9. doi: 10.1515/CCLM.2006.123. PMID 16729864
- [Background] Maheu-Cadotte, M., et al. (2020). Designing effective educational games for nursing education. Nurse Education Today, 92, 104490.
- [Background] Luctkar-Flude, M., et al. (2021). Virtual simulation in nursing education: A systematic review. Journal of Nursing Education, 60(6), 319-325.
- [Background] Keys, M. D., et al. (2020). Simulation in nursing education: An integrative review. Nursing Education Perspectives, 41(2), 83-89.
- [Background] Green, S. F. (2013). The cost of preanalytical errors. Clinical Laboratory News, 39(5), 1-5.
- [Background] Foronda, C. (2021). The effectiveness of virtual simulation in nursing education. Nurse Educator, 46(3), 124-130.
- [Background] Alcantara, C. S., et al. (2022). Preanalytical errors in venous blood sampling. Journal of Clinical Pathology, 75(4), 217-224.